# **Study Protocol**

Title: A Randomized Controlled Trial on the Application of Artificial Intelligence (AI) in Skin Assessment for Pressure Injury Prevention and Staging by Critical Care Nurses

NCT Number: Not Available as yet

Document Date
December 5, 2025



مستشفى الملك فيصل التخصصي ومركز الأبحاث King Faisal Specialist Hospital & Research Centre مؤسسة عامة . Gen. Org. فرع جدة - Jeddah Branch

# Institutional Review Board (IRB)

# **Application for Approval** of Research Proposal

# **RESEARCH PROPOSAL PACKAGE**

# **CONTENTS:**

- 1. COVER SHEET
- 2. DEPARTMENTAL APPROVAL FORM
- 3. ABSTRACT
- 4. PROPOSAL
- 5. WORK PLAN & RESPONSIBILITIES
- 6. REFERENCES
- 7. BUDGET SHEET
- 8. PHARMACY INFORMATION SHEET
- 9. BIOLOGICAL HAZARDS FORM
- 10. INFORMED CONSENT FORM [KFSH&RC(Gen.Org.)-Jeddah Branch Format]
- 11. CASE REPORT FORM

ANNEX A. CURRICULUM VITAE OF PRINCIPAL INVESTIGATORS

ANNEX B. HUMAN PARTICIPANT PROTECTIONS EDUCATION FOR RESEARCH TEAMS COMPLETION CERTIFICATE

(FOR RESEARCHERS WHO HAVE NO PUBLISHED RESEARCH PAPERS YET)

FOR COLLABORATIVE STUDIES /INDUSTRY STUDIES (COMPANY SPONSORED)

ANNEX C. PROTOCOL / INFORMED CONSENT

ANNEX D. CASE REPORT FORM(S) / QUESTIONNAIRE

ANNEX E. SERIOUS ADVERSE EVENTS (FOR INDUSTRY STUDIES ONLY)

ANNEX F. INVESTIGATOR'S BROCHURE (FOR INDUSTRY STUDIES ONLY)

| No. |
|------------------|
| Submission Date: |

# 1. IRB RESEARCH PROPOSAL - COVER PAGE

| Title of Proposal: A Randomized Controlled Trial on the Application of Artificial | Duration of Study: |
|---|---|
| Intelligence (AI) in Skin Assessment for Pressure Injury Prevention and Staging by Critical | |
| Care Nurses | |

# 2. DEPARTMENTAL APPROVAL

<u>Title of Proposal</u>: A Randomized Controlled Trial on the Application of Artificial Intelligence (AI) in Skin Assessment for Pressure Injury Prevention and Staging by Critical Care Nurses

# **Approval - Departmental Research Committee:**

The Committee has reviewed this proposal and attests to its scientific validity.

| Departmental Research Committee Designee | Signature | Date |
|------------------------------------------|-----------|------|

# **Approval - Department Head(s):**

I have reviewed this proposal and approve the participation of the concerned personnel of my department in it.

| PARTICIPANTS | DEPARTMENTAL CHAIRMAN<br>/UNIT HEAD | SIGNATURE |
|--------------|-------------------------------------|-----------|
| | | WE I |

### **Declaration of Conflict of Interest:**

All investigators must declare <u>any</u> potential conflict of interest with respect to this research proposal. The presence of such conflict of interest must be explained (see below). The lack of such declaration by investigators involved with this proposal is taken as evidence of the absence of any conflict of interest.

#### **Conflict of Interest:**

| NAME | SIGNATURE | EXPLANATION |
|------|-----------|-------------|

# 3. ABSTRACT

Should not exceed 200 words and should include:

- The importance of the research topic
- The research hypothesis, question or statement, specific objectives and the significance of the outcome
- OUTLINE the methods that will be used to accomplish the research specific objectives

# **Background**

Pressure injuries are a common issue in healthcare, especially in ICU patients due to immobility and critical conditions. Traditional skin assessments by nurses are effective but vary due to differences in skill and experience. This variability can impact early detection of pressure injuries. Using artificial intelligence (AI) in skin assessment offers promise by utilizing image recognition to identify high-risk patients, monitor skin changes, and suggest timely interventions.

#### Aim

The aim of this study is to examine the effectiveness and impact of Al-assisted skin assessments and Pl staging in critical care settings, by comparing its accuracy, reliability, and nurses' confidence and knowledge with those of traditional assessment methods employed by critical care nurses.

#### Methods

Experimental Research design, with a control and Intervention group will be followed. The setting will include the medical intensive care unit. Critical care nurses (91) will be randomized. Pre and post intervention data on the knowledge and confidence re skin assessment and pressure injury staging will be collected using **Principal Investigator:** 

| Name (print) | Signature: | Date: |
|--------------|------------|-------|

tools that will be piloted. Control group nurses will assess the skin using standard self-assessment techniques, whilst the nurses in the intervention group will use an artificial intelligence app. A senior wound care expert will complete a third assessment which will form part of the verification process. The National Pressure Injury advisory Panel gudielesmes will be used for the assessment. Patients will be consent solely for the purpose of the skin assessment.

#### Conclusion

Understanding the burden of pressure injuries in ICU settings has prompted researchers and clinicians to explore innovative approaches for early detection and informed assessment

# Keywords

Artificial intelligence, critical care, intensive care, nurses, pressure injurie

# 4. RESEARCH PROPOSAL

**Title of Proposal:** A Randomized Controlled Trial on the Application of Artificial Intelligence (AI) in Skin Assessment for Pressure Injury Prevention and Staging by Critical Care Nurses

#### Introduction

May include background information related to the research topic (Importance of the topic), the purpose in carrying out this research, and the importance of potential (expected) findings.

# **Background**

Pressure injuries (PIs) are among the most prevalent issues encountered worldwide in healthcare settings (Feuchtinger et al., 2007), yet they are largely preventable (Slawomirski et al., 2017). A meta-analysis estimates the global incidence of hospital-acquired pressure injuries at about 5.4 per 10,000 hospital patients per day (Li et al., 2020). While the global prevalence of pressure injuries in hospitalized adults is around 12% (Li et al., 2020; Rodgers et al., 2021), the prevalence of hospital-acquired pressure injuries typically ranges from 7% to 9% (Li et al., 2020; Rodgers et al., 2021). These injuries can lead to extended hospital stays, increased healthcare costs, and severely affect patient outcomes, leading to complications such as infections and prolonged pain (Gorecki et al., 2009). Resources required to treat PIs, including nursing time and incremental wound care costs, significantly burden healthcare systems. Treating broken skin PIs can cost healthcare organizations between \$20,900 and \$151,700 per injury (Bouyer-Ferullo et al., 2021). The

annual treatment costs to the US healthcare system associated with hospital-acquired pressure injuries (HAPIs) exceed \$27 billion (Padula & Delarmente, 2019).

PIs are preventable complications acquired in healthcare settings (European Pressure Ulcer Advisory Panel et al., 2019) and are influenced by the quality of nursing care (Burston et al., 2014; Sim et al., 2018; Twigg et al., 2019). These injuries result in unnecessary harm, including pain, psychological distress, reduced quality of life, and, in severe cases, death (Gorecki et al., 2012; Jackson et al., 2017; Jackson et al., 2018; Kim et al., 2019). As a result, healthcare professionals, researchers, and safety experts have focused on strategies to prevent them. Numerous approaches to risk assessment and prevention have been explored (Beeckman et al., 2021; Lovegrove et al., 2021; McLaren-Kennedy et al., 2023). However, pressure injuries still affect approximately 8% of hospitalized patients (Li et al., 2020), with rates being higher in specific highrisk groups, such as the elderly (Rasero et al., 2015), critically ill patients (Labeau et al., 2021), and those with spinal cord injuries (Shiferaw et al., 2020).

ICU patients are particularly vulnerable to PIs due to their immobility and the critical nature of their health conditions (Jacq et al., 2021). The development of PIs in ICUs is a complex, multifactorial process that can be difficult to prevent (Labeau et al., 2021). Contributing factors such as neurological impairments, life-saving medical treatments, fluid resuscitation, vasoactive medications, and pathophysiological conditions that hinder repositioning all increase the risk of PI formation in ICU patients (Gefen et al., 2021). As a result, ICUs experience a higher incidence of PIs compared to other healthcare environments, placing significant physical, psychological, and financial strain on patients who are among the most critically ill in the healthcare system (Chaboyer et al., 2018).

Preventing HAPIs is a critical aspect of patient safety and quality of care, and is often considered an indicator of nursing care quality, as nurses are primarily responsible for assessing patients' risk for PIs and managing skin integrity. While prevalence is not an absolute measure, it serves as an outcome indicator (rather than a process measure) to reflect the quality of care provided. Previous research has indicated that nurses' knowledge of skin assessment, PI risk factors, and positive attitude toward prevention measures play key roles in reducing the incidence of PIs (Taliier et al., 2027).

However, research also indicates that nurses' knowledge about the prevention and treatment of pressure injuries (PIs) is not optimal. For instance, Gunningberg and colleagues (2012) assessed 415 healthcare professionals in Sweden (including RNs, nursing assistants, and student nurses) and found a mean score **Principal Investigator:** 

| Name (print) | Signature: | Date: |
|--------------|------------|-------|

of 58.9% on a test designed to evaluate PI prevention knowledge. Similarly, Karabag Aydin and Karadag (2013) studied 237 nurses in Turkey on their understanding and practices regarding deep tissue injury and stage 1 PIs, revealing a mean score of 48.85 out of 100. Sving and colleagues (2014) conducted a 1-day prevalence study involving 825 patients in both a university-based and community-based hospital in Sweden. They found that preventive interventions were implemented in 44.1% to 58.7% of patients at risk for PIs. A recent survey of 347 nurses attending the 2013 and 2015 Wound Management Congresses found a mean score of 57.37  $\pm$  14.26 out of 100 on 27 items related to pressure injury knowledge and practices (Aydin et al., 2019).

Further, literature reveals limited evidence regarding the accuracy of nurses' skills and knowledge in PIs staging and documentation. A 2012 wound care study found that only 55% of 647 nurses could correctly identify the stages of PIs in their patients. Additionally, just 32% of respondents reported receiving adequate education on chronic wounds during their basic nursing training. In a quality improvement initiative led by Dahlstrom et al., aimed at enhancing the identification, documentation, and treatment of PIs, complete documentation (including stage, size, and location) improved from 29% to 46% after implementing a wound assessment form and point-of-care reminders. However, despite this improvement, more than 50% of the documented injuries were inaccurately recorded. These findings highlight ongoing challenges with nurses' ability to accurately stage and document pressure injuries.

Further, nurses' confidence in conducting skin assessments plays a crucial role in the early detection and prevention of pressure injuries (PIs). Studies show that confidence in performing skin assessments positively impacts nurses' ability to identify pressure injuries early and implement effective preventive strategies. For instance, when nurses feel confident in their skills, they are more likely to conduct thorough assessments and take timely actions to prevent pressure injuries (Stechmiller et al., 2011). Conversely, lack of confidence can lead to missed detections, delayed interventions, and increased risk of complications for patients (Bergstrom et al., 2019). Training and continuous education are key to enhancing nurses' confidence in skin assessment, ensuring that they feel capable of using assessment tools and applying clinical judgment accurately (Coleman et al., 2017). Furthermore, improved confidence has been linked to better patient outcomes, as nurses are more likely to engage in preventive measures such as repositioning and using pressure-relieving devices (Tawfik et al., 2020).

Preventing pressure ulcers has been a longstanding nursing concern, with Florence Nightingale noting in 1859 that bedsores were often a result of poor nursing rather than the disease itself (Nightingale, 1859). **Principal Investigator:** 

| Name (print) | Signature: | Date: |
|--------------|------------|-------|

While some attribute pressure ulcer development to inadequate nursing care, many clinicians see it as a systemic failure involving the entire healthcare team, including nurses, physicians, physical therapists, and dietitians (AHRQ, 1992). Despite being a multidisciplinary responsibility, nurses play a major role in prevention. The 1992 guidelines from the U.S. Agency for Healthcare Research and Quality (AHRQ) continue to serve as a foundational resource for pressure ulcer prevention, highlighting key processes such as risk assessment, skin care, and patient education (AHRQ, 1992).

Comprehensive skin assessments are essential for identifying early skin changes, which can contribute significantly to preventing PIs (Mitchell, 2018; Shi et al., 2018). These assessments provide an opportunity to reposition patients, educate them about skin health, and implement protective measures (Moore & Paton, 2019). Several studies indicate that frequent comprehensive skin assessments can reduce the risk of developing PIs (Fischbein, 2023; Moore & Paton, 2019; Mitchell, 2018; Shi et al., 2018; Coleman et al., 2018; Hommel et al., 2017; Coyer et al., 2017; Reddy et al., 2006).

The National Pressure Injury Advisory Panel (NPIAP) staging system is a widely used framework for classifying the severity of PIs. This system helps healthcare professionals assess and document the extent of tissue damage in patients with pressure injuries, guiding treatment and management decisions. The NPIAP staging system classifies pressure injuries based on the severity of tissue damage. It includes Stage I, characterized by non-blanchable redness of intact skin, Stage II, involving partial-thickness loss of skin, Stage III, with full-thickness skin loss potentially extending into subcutaneous tissue, and Stage IV, where there is extensive damage to deeper structures like muscle or bone. The system also includes unstageable, where necrotic tissue, and Deep Tissue Pressure Injury (DTPI), marked by deep, non-blanchable discoloration or a blood-filled blister, obscure the depth. These stages help guide the assessment, treatment, and prevention of pressure injuries in clinical settings. (National Pressure Injury Advisory Panel, 2016).

Accurate staging of PIs is essential for effective nursing care management (García-Fernández, et al, 2014). However, other skin conditions, such as friction injuries, moisture-associated skin damage (MASD), incontinence-associated skin damage (IAD), and mixed-etiology wounds, which also cause skin inflammation, may present similarly to PIs, resulting in incorrect staging. This misclassification can lead to inappropriate treatment, especially in the case of MASD, which is often mistaken for stage 1 or 2 PIs (Beeckman et al, 2007; Ham et al, 2025).

| Name (print) | Signature: | Date: |
|-------------------------------------------|------------|-------|
| Problem Statement Principal Investigator: | | |

Pressure injuries represent a significant clinical challenge within the ICUs where patients are often immobilized, have compromised skin integrity, and face numerous other health risks. These injuries can lead to extended hospital stays, increased healthcare costs, and severely affect patient outcomes, causing complications such as infections and prolonged pain (Gorecki et al., 2009). Despite existing preventive measures, hospital-acquired pressure injuries (HAPIs) remain prevalent, particularly among vulnerable populations like critically ill ICU patients who face additional challenges in preventing these injuries due to their complex medical needs. Furthermore, despite advancements in PI prevention protocols, the knowledge gap among healthcare professionals about PI risk factors, staging, and prevention strategies still exists, contributing to suboptimal outcomes. This highlights the need for continuous education and improved clinical practices to reduce the incidence of pressure injuries in healthcare settings.

Understanding the burden of pressure injuries in ICU settings has prompted researchers and clinicians to explore innovative approaches for early detection and informed assessment. Traditional methods of skin assessment, typically performed by nurses, have proven effective but are subject to variability in skill and experience among nursing staff. This variability can impact the accuracy of detecting early-stage pressure injuries, highlighting the need for more reliable assessment techniques (Labeau et al, 2021). Implementing artificial intelligence (AI) as a tool to assist in skin assessment and staging of pressure injuries holds great promise in addressing this challenge. Al-driven technologies, such as image recognition, can support clinical decision-making by identifying high-risk patients, monitoring changes in skin integrity, and recommending appropriate interventions in real time. By integrating AI into pressure injury prevention and management strategies, hospitals can improve patient outcomes, reduce the incidence and severity of HAPIs, and optimize resource utilization. Furthermore, AI can standardize wound care approaches, ensuring consistency in both assessment and nursing documentation. Ultimately, the integration of AI into these strategies can enhance patient safety and improve overall healthcare efficiency (Dweekat et al, 2024).

As of March 2025, Al tools for pressure injury assessment are gaining traction in healthcare settings due to their potential to improve patient care and clinical efficiency. Al models have demonstrated significant improvements in accuracy and efficiency, with deep learning-based models achieving 74% Intersection over Union (IoU) and 83% accuracy for wound bed segmentation, outperforming the Braden Scale's 54% accuracy (Keller, 2024). These tools also save time, with Al systems reducing wound assessment time and potentially saving up to 250 labor hours per day in a 500-bed facility (Keller, 2024). Additionally, predictive **Principal Investigator:** 

| Name (print) | Signature: | Date: |
|-----------------|------------|--------|
| realite (princ) | | Dutter |

Al models have shown a 20% improvement in predicting patients at risk of pressure injuries, with an accuracy of over 74% (Keller, 2024). Despite not being universally adopted, Al adoption is expanding, with hospitals and research institutions actively developing Al-powered systems (Liu et al., 2025; Keller, 2024; Alderden et al., 2024). The Al wound care market is projected to grow from \$3.32 billion in 2025 to \$7.65 billion by 2030 (Kronikare, 2025). However, challenges remain in integrating Al tools, including data privacy, algorithm training, and equitable access (Liu et al., 2025; Keller, 2024).

# AT THE CURRENT INSTITUTION, WITHIN THE CRITICAL/INTENSIVE CARE UNITS

As illustrated in Figure 1, the organization recorded 150 cases of stage two and above HAPIs in 2024. Of these, 76 cases (51%) occurred in the critical care setting. The cost for a one-day stay in the MSICU is 8,300 SR, excluding additional procedures. The cost of wound or pressure injury dressings varies depending on the consumables used for each patient. However, based on the average cost for a medium-sized dressing with twice-daily changes, the daily cost per patient is approximately 200 SR.



Figure 1: Total HAPIs for 2024

| Principal Investigator: | | |
|-------------------------|------------|-------|
| Name (print) | Signature: | Date: |

# **Conceptual Framework**

This study will be guided by the Donabedian's Model of Quality Care which focuses on three key components: structure, process, and outcome:

This model emphasizes that high-quality healthcare requires optimal structure, effective processes, and positive outcomes, providing a comprehensive approach for evaluating and improving healthcare services.

#### **STRUCTURE**

Attributes of the settings where care takes place, including the physical facilities, resources, and the personnel involved in care

#### **PROCESS**

Involves how healthcare is delivered, focusing on the interactions between healthcare providers and patients, and the actual delivery of care

#### **OUTCOME**

Refers to the results of healthcare services, such as improvements in patient health, satisfaction, and the overall effectiveness of care

1

1

- Personnel: The study will involve critical care nurses with training in Al skin assessment technology.
- Technology: Al-based skin assessment tools, which might include image recognition software or sensor-based systems that identify early signs of pressure injuries.
- Environment: The study will be conducted in critical care units, where patients are at high risk for pressure injuries.
- Protocols: Standardized pressure injury prevention protocols will be integrated with Al tools such as the NPIAP quidelines.

- Skin Assessment
  Process: The systematic
  - use of Al by critical care nurses to assess patients' skin for early signs of pressure injuries and staging thereof. This could include nurses using Al to scan the skin, interpret results, and document findings.
- **Decision-Making:** Nurses use Al-generated insights (e.g., early detection of pressure injuries or skin breakdown) to make decisions about interventions like repositioning, wound care, using preventive measures such as special mattresses.
- Collaboration with Other Healthcare Providers: How nurses work with other team members (e.g., wound care specialists, doctors) to ensure that AI findings are discussed and acted upon in the context of patient care.

Al Accuracy: The study would analyze accuracy of the Al in detecting early pressure injuries compared to standard clinical methods.

1

- Nurses' confidence: The study will measure whether nurses feel more confident when using AI technology for skin assessments
- Nurses' knowledge:. The study will measure whether nurses feel more knowledgeable when using Al technology for skin assessments as opposed to the traditional methods.

| Figure 2: Donedebian's Framework of | Quality Care (Donabedian,1988) | ) |
|---|---|---|
| Aim | | |
| The aim of this study is to examine to staging in critical care settings, by commute the with those of traditional assessment means to the study is to examine the staging in critical care settings, by commute the study is to examine the staging in critical care settings, by commute the study is to examine the staging in critical care settings. | paring its accuracy, reliability, an | d nurses' confidence and knowledge |
| Objectives | | |
| standard assessments by critic | cal care nurses.<br>nd confidence in using Al for skin | ents and PI staging in comparison to assessment and PI staging versus |
| Research Hypothesis | | |
| Al-assisted skin assessments and pre compared to standard assessments by | | rate greater accuracy and reliability |
| Principal Investigator: | | |
| Name (print) | Signature: | Date: |

## Methodology

May include: 1. Inclusion Criteria and Exclusion Criteria, which will be used in selecting the research participants; 2. Registration, 3. Randomization Process, 4. Data gathering methods, 5. Procedures, Designated Central Laboratories, 6. Follow-up, 7. Safety and Efficacy Parameters, 8. Expected Outcome, 9. Sample Size, and 10. Statistical Methods.

| Methodolog | ٧ | oa | olo | od | th | e | M |
|------------|---|----|-----|----|----|---|---|
|------------|---|----|-----|----|----|---|---|

Research Design

The study will follow a basic experimental research design- pre post-test design.

# Research Setting

The research setting will include the Medical Surgical Intensive Care (MSICU) at King Faisal Specialist Hospital and Research- Center- Jeddah. MSICU is an 18-bedded unit, which houses patients who are requiring intensive care for conditions such as:

- All critically ill Medical patients requiring intensive care or observation.
- Respiratory failure, cardiac failure, liver failure and/or renal failure.
- Critically ill Hematology/Oncology, Immuno-compromised patients.
- •Shock (Cardiogenic, Septic, Anaphylactic, Neurogenic).
- Neurological cases ischemic or hemorrhagic pathologies

# Population

The study will include critical care nurses. Table 1 below provides information re the breakdown of the total number of nurses:

| Job Title | Occupied |
|-------------------------|----------|
| STAFF NURSE III | 2 |
| Principal Investigator: | |

Signature:

Date:

Name (print)

| STAFF NURSE I | 86 |
|-----------------|----|
| NURSE CLINICIAN | 1 |
| NURSE CLINICIAN | 1 |
| Total | 90 |

Sampling technique and sample size:

All critical care nurses who are eligible and who consent to participate will be included for a possible total of up to n=90. The study will focus on one ICU initially (the MSICU) to assess feasibility of the proposed methods. A simple random sampling approach will be followed for allocation into the control (n=45) and intervention group (n-46).

#### Inclusion criteria

- Nurses working within the organisation for at least 6 months
- Nurses involved in direct patient care for over 50% of their work time.
- Skin assessments and staging for patients at risk for developing pressure injuries (Using the Braden Scoring system).
- Adult Patients (18 years and older)
- Patients who are currently admitted to the ICU and are receiving critical care treatment.
- No current severe skin conditions patients without active severe dermatological conditions (e.g., large open wounds, severe rashes) that would interfere with the Al-based skin assessment process.

### Exclusion criteria

- Nurses working within the organization for less than 6 months
- Nurses involved in direct patient care for less than 50% of their work time
- End-of-Life Care or Terminal Illness- patients receiving end-of-life care or those with a terminal diagnosis, where the prevention of pressure injuries may not be a priority and where participation in the study may not align with their care goals.

| Principal Investigator: | | |
|-------------------------|------------|-------|
| Name (print) | Signature: | Date: |

- Severe or active dermatological conditions- patients with active skin conditions such as severe rashes, burns, or other dermatological issues that could interfere with accurate skin assessments by AI or confound the study results.
- Recent Skin Grafts or Advanced Wound Care- patients who have recently undergone skin grafts or those receiving complex wound care treatments that are outside the scope of typical pressure injury prevention practices.
- Inability to Maintain Required Positioning for Skin Assessment- patients who are physically unable to remain in the necessary position for the skin assessments, either due to severe mobility restrictions or critical medical conditions.

# **Current practice**

At KFSHRC, nursing staff in critical care areas follow a standardized skin assessment protocol aligned with the National Pressure Injury Advisory Panel (NPIAP) standards for pressure injury prevention, as outlined in hospital policy (CIPP-3818: Pressure Injury Prevention and Skin Integrity Maintenance). A comprehensive head-to-toe skin assessment is conducted within the first two hours of patient's admission, transfer, or the beginning of each shift, using visual inspection to evaluate skin integrity and identify early signs of pressure injuries. The Braden Scale, a validated tool for pressure injury risk assessment, is used for all patients aged 18 years and older. A Braden score of ≤18 indicates increased risk, requiring appropriate preventive measures. High-risk areas, including the sacrum, buttocks, heels, occipital region, and elbows, receive special attention during assessments. For patients identified as at risk, skin assessments are performed at least every two hours during repositioning, in addition to a daily pressure injury risk assessment documented in the Integrated Clinical Information System (ICIS). The frequency of assessments is increased in response to clinical deterioration or newly identified risk factors, such as hemodynamic instability, impaired mobility, moisture-associated skin damage, decreased perfusion, or compromised nutritional status. If a pressure injury is identified, it is documented in ICIS, and patients with Stage 2 or higher injuries are referred to the Wound Care Specialist or Nurse champion for further evaluation, staging, and treatment recommendations. By adhering to the evidence-based hospital protocols, this systematic approach ensures early detection of pressure injury risk and timely implementation of preventive interventions, promoting patient safety and skin integrity in critical care settings.

| Principal Investigator: | | |
|-------------------------|------------|-------|
| Name (print) | Signature: | Date: |

# Intervention - See below flo



| Feature | Control Group (Manual) | Intervention Group (Al- |
|-------------------|----------------------------|--------------------------|
| | Assessment | Assisted) |
| Technology use | None | Al software (Mobile app) |
| Training required | Standard skin assessment | Nursing trained on using |
| | and staging training as | Al tool |
| | indicated above | |
| Accuracy of | Manual Inspection by nurse | Al Assisted assessment |
| assessment | | based in Al visual data |
| | | analysis |
| Decision support | Nurses clinical judgement | Al Alerts and |

Wound Care Specialist Expert review

Name (print)

**Principal Inve** 

Post-Intervention assessment:

Knowledge and confidence skin assessment and staging OX Comparison of accuracy of Assessment by O and X

Research Proposal Application Form Institutional Review Board- KFSH&RC-Jeddah IRB Forms – Revised on 26 September 2017

Data analysis

# Expert assessment:

In this randomized controlled trial, the wound care expert responsible for evaluating the outcomes will be blinded to the study group assignments to prevent any potential bias. The expert will independently assess the skin, which will be de-identified and presented without any information regarding whether the assessments were conducted using the AI tool or through traditional methods by the critical care nurses. This ensures that the wound care expert's evaluation is based solely on the clinical characteristics of the skin, without influence from the method of assessment. By performing her own independent assessment, the expert maintains objectivity, allowing for an unbiased comparison of the nurses in the intervention and control group in pressure injury prevention.

#### Pre-education on skin assessment

- 1. To enhance nurses' proficiency in using a structured risk assessment approach—such as the Braden Scale—within 2 hours of admission, every 12 hours, or upon a change in condition, considering additional risk factors, and implementing individualized care plans based on the overall risk assessment and Braden subscales to effectively prevent pressure injuries.
- 2. To equip nurses with the skills to perform comprehensive skin assessments—using visual inspection and palpation—upon admission, transfer, and every shift, focusing on identifying erythema, discoloration, edema, and temperature changes across all bony prominences and during every patient turning, ensuring timely interventions and accurate documentation for pressure injury prevention.
- To equip nurses with the skills to perform specialized skin assessments for diverse patient
  populations, including techniques for assessing patients with dark skin tones, monitoring skin under
  medical devices, confidently staging pressure injuries, and ensuring timely interventions for pressure
  injury prevention.
- 4. To enhance critical care nurses' knowledge and skills in utilizing Artificial Intelligence (AI) tools for accurate skin assessment, early detection, accurate staging, and effective prevention of pressure injuries.

| Principal Investigator: |
|-------------------------|

Choice of Artificial Intelligence Tool:

ChatGPT will be utilized in this research project specifically to assist in the skin assessment of the intervention group, where critical care nurses will use AI tools to evaluate pressure injuries based on the National Pressure Injury Advisory Panel (NPIAP) guidelines. The NPIAP guidelines provide a standardized approach to assessing pressure injuries, including identifying stages of injury, determining tissue damage, and evaluating risk factors. ChatGPT will assist in reviewing and synthesizing the NPIAP guidelines to ensure that the AI tool is being used in alignment with current best practices for pressure injury assessment. The model will also help analyze the AI-assisted skin assessment results, comparing them to NPIAP standards to evaluate the tool's accuracy in identifying the severity of pressure injuries, determining the

proper staging, and ensuring proper documentation of skin conditions. By using ChatGPT, the research

team can efficiently analyze the Al's effectiveness in applying NPIAP criteria for accurate and consistent skin assessments

To standardize the use of cameras in the current research study particularly when using the camera for image capturing consistent camera specifications such as, lighting, and positioning will be maintained. Different phone models will be used, hence their performance will be tested to ensure consistency. Photos will be taken under controlled lighting conditions, with established positioning guidelines to maintain the same distance, angle, and orientation for each shot, potentially using a tripod or stand for consistency. Additionally, a standardized camera app will be used across all devices to ensure uniform settings. Training for all personnel involved in the study is essential to ensure adherence to protocols, and regular testing and validation of images will be conducted to ensure quality is maintained. Clear protocols for storing and labeling images will be used and is necessary for proper tracking and analysis for the use of the AI. The study team will ensure that at least three cellphones will be provided to the unit, to avoid any personal cellphones being

Data collection

| Data | will | he | col | lected | hv. |
|------|-------|----|-----|--------|-----|
| Data | AAIII | | CUI | 16666 | DV. |

1. A questionnaire:

Section 1: Demographic section of participants

used so that personal phones are not used.

**Principal Investigator:** 

| Name (print) | Signature: | Date: |
|--------------|------------|-------|

Section 2; The Pressure Ulcer Prevention Knowledge Assessment Instrument (PUPKAI) is a tool designed to assess knowledge on preventing and recognizing pressure ulcers through multiple-choice questions. It can be used in a self-report or interview format and consists of 26 items organized into six themes: Aetiology and Development (6 items), Classification and Monitoring (5 items), Risk Assessment (2 items), Nutrition (1 item), Preventive Interventions to reduce pressure/shear (7 items), and Preventive Measures to reduce pressure duration (5 items). Each item has three response options, with one correct answer. The highest possible score is 26, and a score of 16 (60%) is considered proficient (Beeckman, et

The psychometric properties of PUPKAI have been evaluated. Beekman et al (2010) reported good internal consistency (Cronbach's alpha = 0.77) and strong test-retest reliability (intra-class correlation = 0.88). The content validity index ranged from 0.78 to 1.0. However, differences were noted in the test's performance across different groups, indicating variations in known-groups validity. Item difficulty ranged from 0.27 to 0.87, and discrimination values ranged from 0.29 to 0.65. The original version has been widely used in studies (Shouli et al, 2024; Dirgar et al, 2022; Liu et al, 2017).

Section 3: **Skin Assessment Confidence Scale (SACS)** is a tool designed to assess the confidence levels of nurses in performing skin assessments related to pressure injury prevention. It provides a structured way to measure nurses' self-reported confidence in various key tasks such as identifying early signs of pressure injury, using risk assessment tools, recognizing different stages of pressure injury, and implementing preventative measures. Each item is rated on a 5-point scale (1 = Not Confident, 5 = Very Confident), with a total score that reflects overall confidence. Scores range from 10 to 50, with higher scores indicating greater confidence:

- Total Confidence Score: Add the scores for all 10 questions.
- o 10-20: Low Confidence

al, 2010)

- o 21-30: Moderate Confidence
- o 31-40: High Confidence
- o 41-50: Very High Confidence

The SACS was self-developed and will be piloted with nurses from other intensive care areas namely SCIU, CCU, MICU, SICU-for an acceptable reliability coefficient of ≥.60. In addition, a Test-Retest method will be **Principal Investigator:** 

| Name (print) | Signature: | Date: |
|--------------|------------|-------|

included which will include administering the scale to a group of nurses at two different time points (e.g., one month apart) to assess the stability of the scale over time. A high correlation (e.g., above 0.8) between the two sets of responses would suggest good test-retest reliability. There will be no significant interventions (like training or skill development) take place between the two testing points that might affect participants' responses.

Content validity was ensured by consultation with subject matter experts: Wound Care Specialists, and Wound champions with the current organization who reviewed each item to ensure it accurately reflects the necessary skills and knowledge for skin assessment and pressure injury prevention. These experts were asked to rate each item for relevance to the domain of skin assessment and pressure injury prevention on a Likert scale (e.g., 1 = Not Relevant, 4 = Very Relevant). Items with low relevance scores was revised or removed.

3. Skin Assessment Checklist: NPAIP

See supporting documents attached

#### Data analysis

Continuous variables will be assessed for distribution by comparing median and mean values, by observing skewness, kurtosis, and results from normality tests, and by observing the data graphically. Univariate results will be presented according to distribution of the data as mean ± standard deviation or median (interquartile range) and categorical variables will be represented with frequencies. PUKAT tool results will be scored as previously described (Beeckman, et al, 2010) and SACS will be scored as indicated once scale reliability is confirmed. Bivariable analyses will be used to compare demographics, survey results, and wound assessment between study groups using Chi-square and Fisher's exact tests and Student's t-tests or the non-parametric equivalent as applicable. Agreement between study group assessments and the assessment of the wound care specialist will be analyzed using interrater reliability and Kappa statistics. Survey results from pre and post the education assessment will also be compared using correlation analysis and/or paired t-tests for results within study groups and independent sample t-tests between study groups

| Name (print) | Signature: | Date: |
|-------------------------|------------|-------|
| Principal Investigator: | | |
| Ethical considerations | | |

**Patients** 

Even though patients will not be randomized into the control and experimental groups, patients will be

used in the assessments by nurses included in the study.

**Informed Consent:** 

Patients will be provided with clear, comprehensive information about the study, including its purpose, the

use of AI, and potential benefits and risks. They will be informed about their rights to withdraw from the study

at any point without any negative impact on their medical care. For patients who are unable to give consent

(e.g., unconscious or critically ill), a legally authorized representative should be asked to provide consent on

their behalf.

Confidentiality:

All patient data, including Al-assisted skin assessment images and personal health information, will be

kept confidential and stored securely in compliance with hospital policies.

Non-Maleficence (Do No Harm):

The Al system will be tested and proven to be safe, and all care should be provided in a way that prevents

harm. No unnecessary risks should be introduced to patients, and the system should be monitored for any

adverse effects throughout the study.

Justice (Fair Treatment):

Patients must be selected based on clear, appropriate criteria, ensuring that no groups are unfairly

excluded or overrepresented. All patients should have equal access to the benefits of the study, and no

one should be unfairly disadvantaged by the use of AI in skin assessments.

Respect for Autonomy:

Patients will retain their right to make informed decisions regarding their participation. They should

understand that their participation is entirely voluntary and can be withdrawn at any time without affecting

**Principal Investigator:** 

| NI ( | Si | Date |
|--------------|------------|-------|
| Name (print) | Signature: | Date: |

Nurses

**Informed Consent and Autonomy:** 

Nurses involved in the study will receive clear, detailed information about the study's goals, the role of AI in

skin assessments, and the expected outcomes. They should have the opportunity to voluntarily agree to

participate in the study. Like patients, nurses also have the right to withdraw from the study at any time.

**Training and Competence:** 

Nurses will be trained to use the AI system effectively. This includes understanding how to incorporate AI-

driven assessments into their clinical practice, interpreting Al-generated results, and knowing when human

intervention is needed. Ongoing education should be provided to ensure they remain confident and capable

in

Justice (Fair Treatment):

Nurses should be involved in the study equally and fairly, with no discrimination. They should have equal

access to training and resources related to the AI system, ensuring a level playing field across the clinical

team.

**Accountability:** 

Nurses must remain accountable for their actions and decisions when using AI tools. While AI can provide

valuable insights, nurses are responsible for ensuring that the final clinical decisions, particularly in patient

care, are made by considering the full context and not solely relying on Al-generated assessments.

Workload Considerations:

The introduction of AI should not place undue burden on nurses. It is essential that AI tools are designed to

support nurses in their role, reducing workloads where appropriate, and not adding additional complexity or

stress. It is critical that Al tools be implemented in a way that enhances workflow efficiency without

overwhelming staff.

**Principal Investigator:** 

| Name (print) | Signature: | Date: |
|--------------|------------|-------|

# Confidentiality:

No identifying information will be collected for nurses.

# 5. WORK PLAN AND RESPONSIBILITIES

Detailed description of the protocol work plan is mentioned in the original documentation. Please refer to the submitted documents. The following Table summarizes the job responsibilities of involved members:

| Task | Investigator(s) |
|----------------------------------|-----------------|
| Conceptualization of the idea | |
| Writing of the research proposal | |
| Confidence Scale Validation | |
| Accessing IRB Approval | |
| Collection of data | |
| Analysis of the data | |
| Write up of findings | |
| Complete the discussion | |
| Drafting of the manuscript | |

| Principal Investigator: | | |
|-------------------------|------------|-------|
| Name (print) | Signature: | Date: |

# **6. REFERENCES (comprehensive literature review)**

Aydin, A. K., & Karadag, A. (2010). Assessment of nurses' knowledge and practice in prevention and management of deep tissue injury and stage I pressure ulcer. *Journal of Wound Ostomy & Continence Nursing*, 37(5), 487-494.

Aydın, A. K., Karadağ, A., Gül, Ş., Avşar, P., & Baykara, Z. G. (2019). Nurses' knowledge and practices related to pressure injury: a cross-sectional study. *Journal of Wound Ostomy & Continence Nursing*, *46*(2), 117-123.

Beeckman, D., Schoonhoven, L., Fletcher, J., Furtado, K., Gunningberg, L., Heyman, H., ... & Defloor, T. (2007). EPUAP classification system for pressure ulcers: European reliability study. *Journal of advanced nursing*, *60*(6), 682-691.

Beeckman, D., Vanderwee, K., Demarré, L., Paquay, L., Van Hecke, A., & Defloor, T. (2010). Pressure ulcer prevention: development and psychometric validation of a knowledge assessment instrument. *International journal of nursing studies*, *47*(4), 399-410.

Beeckman, D., Fourie, A., Raepsaet, C., Van Damme, N., Manderlier, B., De Meyer, D., ... & Hulstaert, F. (2021). Silicone adhesive multilayer foam dressings as adjuvant prophylactic therapy to prevent hospital-acquired pressure ulcers: a pragmatic noncommercial multicentre randomized open-label parallel-group medical device trial. *British Journal of Dermatology*, *185*(1), 52-61.

| Principal Investigator: | | |
|-------------------------|------------|-------|
| Name (print) | Signature: | Date: |

Bouyer-Ferullo, S., O'Connor, C., Kinnealey, E., Wrigley, P., & Osgood, P. M. (2021). Adding a visual communication tool to the electronic health record to prevent pressure injuries. *AORN journal*, *113*(3), 253-262.

Burston, S., Chaboyer, W., & Gillespie, B. (2014). Nurse-sensitive indicators suitable to reflect nursing care quality: A review and discussion of issues. *Journal of clinical nursing*, *23*(13-14), 1785-1795.

Coleman, S., Smith, I. L., McGinnis, E., Keen, J., Muir, D., Wilson, L., ... & Nixon, J. (2018). Clinical evaluation of a new pressure ulcer risk assessment instrument, the Pressure Ulcer Risk Primary or Secondary Evaluation Tool (PURPOSE T). *Journal of advanced nursing*, 74(2), 407-424.

Chaboyer, W. P., Thalib, L., Harbeck, E. L., Coyer, F. M., Blot, S., Bull, C. F., ... & Lin, F. F. (2018). Incidence and prevalence of pressure injuries in adult intensive care patients: a systematic review and meta-analysis. *Critical care medicine*, *46*(11), e1074-e1081.

Coyer, F., Miles, S., Gosley, S., Fulbrook, P., Sketcher-Baker, K., Cook, J. L., & Whitmore, J. (2017). Pressure injury prevalence in intensive care versus non-intensive care patients: a state-wide comparison. *Australian Critical Care*, *30*(5), 244-250.

Dahlstrom, M., Best, T., Baker, C., Doeing, D., Davis, A., Doty, J., & Arora, V. M. (2011). Improving identification and documentation of pressure ulcers at an urban academic hospital. *The Joint commission Journal on Quality and patient safety*, *37*(3), 123-AP1.

Donabedian, A. (1988). The quality of care: how can it be assessed?. Jama, 260(12), 1743-1748.

Dweekat, O. Y., Lam, S. S., & McGrath, L. (2023). Machine learning techniques, applications, and potential future opportunities in pressure injuries (bedsores) management: a systematic review. *International journal of environmental research and public health*, *20*(1), 796.

| rincipal investigator: |
|-------------------------|
| Principal Investigator: |

Dirgar, E., Tosun, B., Dokumuş, H., & Bülbül, T. (2022). Evaluating nurses' knowledge of pressure injury

prevention: a descriptive study. Advances in Skin & Wound Care, 35(4), 1-6.

European Pressure Ulcer Advisory Panel, National Pressure Injury Advisory Panel, & Alliance, P. P. I.

(2019). Prevention and Treatment of Pressure Ulcers/injuries: Clinical Practice Guideline: The International

Guideline 2019. EPUAP, NPIAP, PPPIA.

Feuchtinger, J., Halfens, R., & Dassen, T. (2007). Pressure ulcer risk assessment immediately after cardiac

surgery-does it make a difference? A comparison of three pressure ulcer risk assessment instruments within

a cardiac surgery population. Nursing in critical care, 12(1), 42-49.

Fischbein, A. B. (2023). Improving skin care protocol use in the intensive care unit to reduce hospital-

acquired pressure injuries. AACN Advanced Critical Care, 34(1), 16-23.

García-Fernández, F. P., Agreda, J. J. S., Verdú, J., & Pancorbo-Hidalgo, P. L. (2014). A new theoretical

model for the development of pressure ulcers and other dependence-related lesions. Journal of Nursing

Scholarship, 46(1), 28-38.

Gefen, A., Brienza, D. M., Cuddigan, J., Haesler, E., & Kottner, J. (2022). Our contemporary understanding

of the aetiology of pressure ulcers/pressure injuries. International wound journal, 19(3), 692-704.

Gorecki, C., Nixon, J., Madill, A., Firth, J., & Brown, J. M. (2012). What influences the impact of pressure

ulcers on health-related quality of life? A qualitative patient-focused exploration of contributory factors.

Journal of tissue viability, 21(1), 3-12.

**Principal Investigator:** 

Name (print) Signature: \_\_\_\_\_\_ Date: \_\_\_\_\_

Gunningberg, L., Mårtensson, G., Mamhidir, A. G., Florin, J., Muntlin Athlin, Å., & Bååth, C. (2015). Pressure ulcer knowledge of registered nurses, assistant nurses and student nurses: a descriptive, comparative multicentre study in Sweden. *International wound journal*, 12(4), 462-468.

Ham, W. H., Schoonhoven, L., Schuurmans, M. J., Veugelers, R., & Leenen, L. P. (2015). Pressure ulcer education improves interrater reliability, identification, and classification skills by emergency nurses and physicians. *Journal of emergency nursing*, *41*(1), 43-51.

Hommel, A., Gunningberg, L., Idvall, E., & Bååth, C. (2017). Successful factors to prevent pressure ulcers—an interview study. *Journal of Clinical nursing*, *26*(1-2), 182-189.

Jacq, G., Valera, S., Muller, G., Decormeille, G., Youssoufa, A., Poiroux, L., ... & Michel, P. (2021). Prevalence of pressure injuries among critically ill patients and factors associated with their occurrence in the intensive care unit: The PRESSURE study. *Australian Critical Care*, *34*(5), 411-418.

Jackson, D., Durrant, L., Bishop, E., Walthall, H., Betteridge, R., Gardner, S., ... & Usher, K. (2017). Pain associated with pressure injury: a qualitative study of community-based, home-dwelling individuals.

Journal of advanced nursing, 73(12), 3061-3069.

Jackson, D. E., Durrant, L. A., Hutchinson, M., Ballard, C. A., Neville, S., & Usher, K. (2018). Living with multiple losses: insights from patients living with pressure injury. Collegian, 25(4), 409-414.

Kim, J., Lyon, D., Weaver, M. T., Keenan, G., & Chen, X. (2019). The role of psychological distress in the relationship between the severity of pressure injury and pain intensity in hospitalized adults. Journal of advanced nursing, 75(6), 1219-1228.

| Principal Investigator: | | |
|-------------------------|------------|-------|
| Name (print) | Signature: | Date: |

Li, Z., Lin, F., Thalib, L., & Chaboyer, W. (2020). Global prevalence and incidence of pressure injuries in hospitalised adult patients: a systematic review and meta-analysis. *International journal of nursing studies*, *105*, 103546.

Labeau, S. O., Afonso, E., Benbenishty, J., Blackwood, B., Boulanger, C., Brett, S. J., ... & DecubICUs Study Team. (2021). Correction to: Prevalence, associated factors and outcomes of pressure injuries in adult intensive care unit patients: the DecubICUs study. Intensive care medicine, 47(4), 503-520.

Lawrence, P., Fulbrook, P., & Miles, S. (2015). A survey of Australian nurses' knowledge of pressure injury/pressure ulcer management. *Journal of Wound Ostomy & Continence Nursing*, 42(5), 450-460.

Lovegrove, J., Fulbrook, P., Miles, S. J., & Steele, M. (2021). Effectiveness of interventions to prevent pressure injury in adults admitted to acute hospital settings: a systematic review and meta-analysis of randomised controlled trials. International journal of nursing studies, 122, 104027.

Liu, M., Yuan, H. B., Chen, W. J., Poon, C., Hsu, M., & Zhang, B. (2016). Translation, modification and validation of the Chinese version of a knowledge assessment instrument regarding pressure ulcer prevention. *Chinese Nursing Research*, *3*(1), 16-23.

McLaren-Kennedy, A., Chaboyer, W., Carlini, J., & Latimer, S. (2023). Use of point-of-care subepidermal moisture devices to detect localised oedema and evaluate pressure injury risk: A scoping review. Journal of Clinical Nursing, 32(17-18), 5478-5492.

Mitchell, A. (2018). Adult pressure area care: preventing pressure ulcers. British Journal of Nursing, 27(18), 1050-1052.

| Principal Investigator: | | |
|-------------------------|------------|-------|
| Name (print) | Signature: | Date: |

Moore, Z. E., & Patton, D. (2019). Risk assessment tools for the prevention of pressure ulcers. *Cochrane Database of Systematic Reviews*, (1).

National Pressure Injury Advisory Panel. (2016). Prevention and Treatment of Pressure Ulcers: Clinical Practice Guideline. Retrieved from <a href="https://www.npiap.com">www.npiap.com</a>.

Padula, W. V., & Delarmente, B. A. (2019). The national cost of hospital-acquired pressure injuries in the United States. *International wound journal*, *16*(3), 634-640.

Rasero, L., Simonetti, M., Falciani, F., Fabbri, C., Collini, F., & Dal Molin, A. (2015). Pressure ulcers in older adults: a prevalence study. *Advances in Skin & Wound Care*, *28*(10), 461-464.

Reddy, M., Gill, S. S., & Rochon, P. A. (2006). Preventing pressure ulcers: a systematic review. *Jama*, *296*(8), 974-984.

Rodgers, K., Sim, J., & Clifton, R. (2021). Systematic review of pressure injury prevalence in Australian and New Zealand hospitals. *Collegian*, *28*(3), 310-323.

Shiferaw, W. S., Akalu, T. Y., Mulugeta, H., & Aynalem, Y. A. (2020). The global burden of pressure ulcers among patients with spinal cord injury: a systematic review and meta-analysis. *BMC musculoskeletal disorders*, *21*, 1-11.

Shouli, M., Bsharat, R., Khalid, H. A., & Shoul, K. (2024). Knowledge and Attitude among Nurses towards Pressure Ulcer Prevention at Palestinian Hospital. *Open Journal of Nursing*, *14*(12), 637-656.

| Name (print) | Signature: | Date: | -000 |
|-------------------------|------------|-------|------|
| Principal Investigator: | | | |

Slawomirski, L., Auraaen, A., & Klazinga, N. (2017). The economics of patient safety. *Paris: Organisation for Economic Co-operation and Development*.

Sim, J., Crookes, P., Walsh, K., & Halcomb, E. (2018). Measuring the outcomes of nursing practice: A Delphi study. *Journal of clinical nursing*, 27(1-2), e368-e378.

Sving, E., Idvall, E., Högberg, H., & Gunningberg, L. (2014). Factors contributing to evidence-based pressure ulcer prevention. A cross-sectional study. *International journal of nursing studies*, *51*(5), 717-725.

Tallier, P. C., Reineke, P. R., Asadoorian, K., Choonoo, J. G., Campo, M., & Malmgreen-Wallen, C. (2017). Perioperative registered nurses knowledge, attitudes, behaviors, and barriers regarding pressure ulcer prevention in perioperative patients. *Applied Nursing Research*, *36*, 106-110.

Twigg, D. E., Kutzer, Y., Jacob, E., & Seaman, K. (2019). A quantitative systematic review of the association between nurse skill mix and nursing-sensitive patient outcomes in the acute care setting. *Journal of advanced nursing*, 75(12), 3404-3423.

| rincipal Investigator: |
|------------------------|

| 7. BUDGET SHEET | | | | | |
|---|---|---|---|---|---|
| PERSONNEL<br>(NAME) | POSITION ON PROJECT | %<br>TIME | GR/STEP | YEAR 1 | YEAR 2 |
| A) total for personnel: | | | | SR | SR |
| EQUIPMENT (use separate shee | t if required) | | | YEA | .R |
| B) total for equipment: | | | | SR | SR |
| SUPPLIES AND MATERIALS (US | se separate sheet if required) | | | YEA | .R |
| C) Total for materials and su | pplies: | | | SR | SR |
| other exper | nses <i>(use separate sheet if r</i> | equired) | | | |
| category | | purpose | | Амоц | JNT |
| D) Total for other expenses: | | | | SR | SR |
| TOTAL BUDGET (A → D) | | | | SR | SR |
| TOTAL BUDGET (A → D) incipal Investigator: | | nature: | | | |

Research Proposal Application Form Institutional Review Board- KFSH&RC-Jeddah IRB Forms – Revised on 26 September 2017

**Suggested Sources of External Funding** Relationship to research proposal **Address Company None** 8. Pharmacy Information Sheet (page 1 of 2) **Title of the Proposal:** IRB #: (if available) \_\_\_\_\_ Principal Investigator: \_\_\_\_ Drug Name Rou EXP Rou EXP Rou EXP Rou EXP Rou EXP Dose Administration Route Administration Frequency Length of Treatment Drug Status\* **Number of Patients** Provider: Hospital or Sponsor (Identify sponsor) **Total Drugs Required** (Pharmacy will calculate) (For Pharmacy Use) Rou Exp Rou Exp Rou Exp Rou Exp Rou Exp medication Cost Research Pharmacist = SR time (hrs) X SR/hr If this is a randomized study, who is responsible for Randomization? Over what period of time do you intend to accrue the patients? The Pharmacy Department must seek approval through the MOH in order to import drugs. Approval of the proposal by the IRB does not guarantee that the drugs will be approved by the MOH. Being a registered or **Principal Investigator:** 

Signature: \_\_\_\_\_ Date:

Research Proposal Application Form Institutional Review Board- KFSH&RC-Jeddah IRB Forms – Revised on 26 September 2017

Name (print)

investigational drug in any of the five reference countries (USA, Canada, UK, Sweden, Saudi Arabia) would help in obtaining MOH approval.

<u>Please use the following abbreviations: **HF** – on Hospital formulary; **MOH** – registered by the Saudi Ministry of Health; **USA** – registered in USA; **CA** – registered in Canada; **UK** – registered in UK; **SW** – registered in Sweden; **USAI** – being investigated in USA; **CAI** – being investigated in UK; **SWI** – being investigated in Sweden.</u>

# PHARMACY INFORMATION SHEET (page 2 of 2)

| (C) | rt is to be completed by the head (*) appropriate box(ex) | he Pharmacy Department: | |
|---|---|---|---|
| | | s) and complete) | |
| | | essigned a Research Pharmacist to prove<br>have any questions, please call the Offi | |
| The<br>I. | Pharmacy department will p<br>Drug keeping and dispensi | | |
| II. | Preparation of Drug | | |
| III. | Drug Information (physicia | | |
| IV. | MOH permit for import, rele | | |
| V. | Patient counseling for drug<br>unused products (if requ | information, compliance, medication haired) | andling, and return of |
| VI. | | s, upon completion/termination of the $s$ $r$ to KFSH&RC: Date, amount, lot $#$ , expressions are $r$ | |
| | (b) use by each stud | y subject | |
| VII. | Follow the trial randomizati | on procedure | |
| VIII | . Supply the drugs listed on I | page 1 of this form | |
| | rmacy Department will be hasfactorily addressed: | ppy to provide the above, provided the | following issues have been |
| 1. | | | |
| 2. | | | |
| 3. | | | |
| ☐ The | Pharmacy Department will r | ot be able to assist with this project du | e to the following: |

| | | | | - | |
|---|---|---|---|---|---|
| | Total Pharmaceutical cost (routi | ine care) | <i>SR</i> Total Pharr | naceutical cost (experimental) | _ SA |
| 9. | BIOLOGICAL HAZAR | DS | | | |
| <u> Fitle c</u> | of the Proposal: | | | | |
| | es the proposed research inv<br>Please name chemicals and | | | ard involved: | |
| 2. | Does the proposed research involve any hazardous micro-organism? If yes, name the organisms and describe the nature of hazards expected. | | | | |
| | Also describe facilities, safet | ty measures and | procedures to | protect personnel and environme | ent. |
| 3. | Does the proposed research If yes, describe the materials, he | | | I personnel protection. | |
| This f | Does the proposed research orm page completed by: | | | | |
| | | | | DATE: | |
| APPR | OVED BY: | SIGN | ATIIPE' | DATE: | |

(Head of Pharmacy Department)

| Describe t | Describe the nature of genes to be cloned, organisms and plasmids to be used. | | |
|---|---|---|---|
| - | | 487. | |
| <b>10. Inforr</b> □ | nformed Consent ☐ for research involving the administration of drugs, use of devices or performance of procedures | | |
| | for research with no | direct benefit to participar | t |
| cipal Investig | ator: | | |
| me (print) | | Signature: | Date: |